CLINICAL TRIAL: NCT01515462
Title: A Phase I/II Clinical Trial of Hematopoietic Stem Cell Gene Therapy for the Wiskott-Aldrich Syndrome
Brief Title: Gene Therapy for Wiskott-Aldrich Syndrome
Acronym: TIGET-WAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Telethon (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201228; 2009-017346-32 (EudraCT Number)
Record Dates: First submitted 2011-12-23; First posted 2012-01-24 (Estimated); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Wiskott-Aldrich Syndrome (WAS)
Keywords: Lentiviral vector; Gene therapy; Wiskott-Aldrich Syndrome; TLT003; Previously GSK2696275; Previously OTL-103
MeSH Terms: conditions — Wiskott-Aldrich Syndrome

STUDY DESIGN:
Intervention Model Description: This will be a single-arm study. All subjects will receive OTL-103 gene therapy and will be followed up for 15 years post gene therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TLT003 gene therapy (Experimental): Eligible subjects will receive intravenous (IV) infusion of TLT003 gene therapy. Subjects affected by WAS who don't have a suitable matched donor for allogenic hematopoietic stem cell transplantation will be included
  Interventions: Genetic: TLT003

INTERVENTIONS:
Genetic: TLT003 — TLT003 is an autologous CD34+ cells collected from bone marrow and/or peripheral blood and transduced with a lentiviral vector encoding Wiskott-Aldrich syndrome (WAS) protein
  Other Names: Previously GSK2696275; Previously OTL-103

SUMMARY:
This is phase I/II protocol to evaluate the safety and efficacy of WAS gene transfer into hematopoietic stem/progenitor cells for the treatment of Wiskott Aldrich Syndrome.

DETAILED DESCRIPTION:
Wiskott-Aldrich Syndrome (WAS) is an X-linked primary immunodeficiency caused by mutations in the WAS gene which encodes the WAS protein (WASP), a cytoskeletal regulator which is expressed exclusively in hematopoietic cells.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of WAS defined by genetic mutation and at least one of the following criteria:

   * Severe WAS mutation
   * Absence of WASP expression
   * Severe clinical score (Zhu clinical score ≥ 3
2. No HLA-identical sibling donor
3. Negative search for a matched unrelated donor (10/10) or an adequate unrelated cord blood donor (5-6/6) within 4-6 months

   * Patients of > 5 years of age who are not candidate to unrelated allogeneic transplant based on clinical conditions.
4. Parental/guardian/patient signed informed consent.

Exclusion Criteria:

1. Patients positive for HIV-infection.
2. Patients affected by neoplasia.
3. Patients with cytogenetic alterations typical of MDS/AML.
4. Patients with end-organ functions or any other severe disease which, in the judgement of the investigator, would make the patient inappropriate for entry into this study.
5. Patients who underwent an allogeneic haematopoietic stem cell transplantation in the previous 6 months.
6. Patients who underwent an allogeneic haematopoietic stem cell transplantation with evidence of residual cells of donor origin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-04-20 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele - Telethon Institute for Gene Therapy (OSR-TIGET), Milan, Italy

REFERENCES:
- [Background] Aiuti A, Biasco L, Scaramuzza S, Ferrua F, Cicalese MP, Baricordi C, Dionisio F, Calabria A, Giannelli S, Castiello MC, Bosticardo M, Evangelio C, Assanelli A, Casiraghi M, Di Nunzio S, Callegaro L, Benati C, Rizzardi P, Pellin D, Di Serio C, Schmidt M, Von Kalle C, Gardner J, Mehta N, Neduva V, Dow DJ, Galy A, Miniero R, Finocchi A, Metin A, Banerjee PP, Orange JS, Galimberti S, Valsecchi MG, Biffi A, Montini E, Villa A, Ciceri F, Roncarolo MG, Naldini L. Lentiviral hematopoietic stem cell gene therapy in patients with Wiskott-Aldrich syndrome. Science. 2013 Aug 23;341(6148):1233151. doi: 10.1126/science.1233151. Epub 2013 Jul 11. PMID 23845947
- [Background] Aiuti A, Cattaneo F, Galimberti S, Benninghoff U, Cassani B, Callegaro L, Scaramuzza S, Andolfi G, Mirolo M, Brigida I, Tabucchi A, Carlucci F, Eibl M, Aker M, Slavin S, Al-Mousa H, Al Ghonaium A, Ferster A, Duppenthaler A, Notarangelo L, Wintergerst U, Buckley RH, Bregni M, Marktel S, Valsecchi MG, Rossi P, Ciceri F, Miniero R, Bordignon C, Roncarolo MG. Gene therapy for immunodeficiency due to adenosine deaminase deficiency. N Engl J Med. 2009 Jan 29;360(5):447-58. doi: 10.1056/NEJMoa0805817. PMID 19179314
- [Background] Aiuti A, Roncarolo MG. Ten years of gene therapy for primary immune deficiencies. Hematology Am Soc Hematol Educ Program. 2009:682-9. doi: 10.1182/asheducation-2009.1.682. PMID 20008254
- [Background] Bosticardo M, Marangoni F, Aiuti A, Villa A, Grazia Roncarolo M. Recent advances in understanding the pathophysiology of Wiskott-Aldrich syndrome. Blood. 2009 Jun 18;113(25):6288-95. doi: 10.1182/blood-2008-12-115253. Epub 2009 Apr 7. PMID 19351959
- [Background] Boztug K, Dewey RA, Klein C. Development of hematopoietic stem cell gene therapy for Wiskott-Aldrich syndrome. Curr Opin Mol Ther. 2006 Oct;8(5):390-5. PMID 17078381
- [Background] Burns S, Cory GO, Vainchenker W, Thrasher AJ. Mechanisms of WASp-mediated hematologic and immunologic disease. Blood. 2004 Dec 1;104(12):3454-62. doi: 10.1182/blood-2004-04-1678. Epub 2004 Aug 12. PMID 15308573
- [Background] Charrier S, Dupre L, Scaramuzza S, Jeanson-Leh L, Blundell MP, Danos O, Cattaneo F, Aiuti A, Eckenberg R, Thrasher AJ, Roncarolo MG, Galy A. Lentiviral vectors targeting WASp expression to hematopoietic cells, efficiently transduce and correct cells from WAS patients. Gene Ther. 2007 Mar;14(5):415-28. doi: 10.1038/sj.gt.3302863. Epub 2006 Oct 19. PMID 17051251
- [Background] Dupre L, Trifari S, Follenzi A, Marangoni F, Lain de Lera T, Bernad A, Martino S, Tsuchiya S, Bordignon C, Naldini L, Aiuti A, Roncarolo MG. Lentiviral vector-mediated gene transfer in T cells from Wiskott-Aldrich syndrome patients leads to functional correction. Mol Ther. 2004 Nov;10(5):903-15. doi: 10.1016/j.ymthe.2004.08.008. PMID 15509508
- [Background] Follenzi A, Sabatino G, Lombardo A, Boccaccio C, Naldini L. Efficient gene delivery and targeted expression to hepatocytes in vivo by improved lentiviral vectors. Hum Gene Ther. 2002 Jan 20;13(2):243-60. doi: 10.1089/10430340252769770. PMID 11812281
- [Background] Galy A, Roncarolo MG, Thrasher AJ. Development of lentiviral gene therapy for Wiskott Aldrich syndrome. Expert Opin Biol Ther. 2008 Feb;8(2):181-90. doi: 10.1517/14712598.8.2.181. PMID 18194074
- [Background] Marangoni F, Bosticardo M, Charrier S, Draghici E, Locci M, Scaramuzza S, Panaroni C, Ponzoni M, Sanvito F, Doglioni C, Liabeuf M, Gjata B, Montus M, Siminovitch K, Aiuti A, Naldini L, Dupre L, Roncarolo MG, Galy A, Villa A. Evidence for long-term efficacy and safety of gene therapy for Wiskott-Aldrich syndrome in preclinical models. Mol Ther. 2009 Jun;17(6):1073-82. doi: 10.1038/mt.2009.31. Epub 2009 Mar 3. PMID 19259069
- [Background] Villa A, Notarangelo L, Macchi P, Mantuano E, Cavagni G, Brugnoni D, Strina D, Patrosso MC, Ramenghi U, Sacco MG, et al. X-linked thrombocytopenia and Wiskott-Aldrich syndrome are allelic diseases with mutations in the WASP gene. Nat Genet. 1995 Apr;9(4):414-7. doi: 10.1038/ng0495-414. PMID 7795648
- [Derived] Quaranta P, Basso-Ricci L, Jofra Hernandez R, Pacini G, Naldini MM, Barcella M, Seffin L, Pais G, Spinozzi G, Benedicenti F, Pietrasanta C, Cheong JG, Ronchi A, Pugni L, Dionisio F, Monti I, Giannelli S, Darin S, Fraschetta F, Barera G, Ferrua F, Calbi V, Ometti M, Di Micco R, Mosca F, Josefowicz SZ, Montini E, Calabria A, Bernardo ME, Cicalese MP, Gentner B, Merelli I, Aiuti A, Scala S. Circulating hematopoietic stem/progenitor cell subsets contribute to human hematopoietic homeostasis. Blood. 2024 May 9;143(19):1937-1952. doi: 10.1182/blood.2023022666. PMID 38446574
- [Derived] Scala S, Ferrua F, Basso-Ricci L, Dionisio F, Omrani M, Quaranta P, Jofra Hernandez R, Del Core L, Benedicenti F, Monti I, Giannelli S, Fraschetta F, Darin S, Albertazzi E, Galimberti S, Montini E, Calabria A, Cicalese MP, Aiuti A. Hematopoietic reconstitution dynamics of mobilized- and bone marrow-derived human hematopoietic stem cells after gene therapy. Nat Commun. 2023 May 27;14(1):3068. doi: 10.1038/s41467-023-38448-y. PMID 37244942
- [Derived] Ferrua F, Cicalese MP, Galimberti S, Giannelli S, Dionisio F, Barzaghi F, Migliavacca M, Bernardo ME, Calbi V, Assanelli AA, Facchini M, Fossati C, Albertazzi E, Scaramuzza S, Brigida I, Scala S, Basso-Ricci L, Pajno R, Casiraghi M, Canarutto D, Salerio FA, Albert MH, Bartoli A, Wolf HM, Fiori R, Silvani P, Gattillo S, Villa A, Biasco L, Dott C, Culme-Seymour EJ, van Rossem K, Atkinson G, Valsecchi MG, Roncarolo MG, Ciceri F, Naldini L, Aiuti A. Lentiviral haemopoietic stem/progenitor cell gene therapy for treatment of Wiskott-Aldrich syndrome: interim results of a non-randomised, open-label, phase 1/2 clinical study. Lancet Haematol. 2019 May;6(5):e239-e253. doi: 10.1016/S2352-3026(19)30021-3. Epub 2019 Apr 10. PMID 30981783

RESULTS

PARTICIPANT FLOW:
Groups:
- OTL-103 Gene Therapy: Eligible subjects will receive intravenous (IV) infusion of OTL-103 gene therapy. Subjects affected by WAS who don't have a suitable matched donor for allogenic hematopoietic stem cell transplantation will be included
  OTL-103: OTL-103 is an autologous CD34+ cells collected from bone marrow and/or peripheral blood and transduced with a lentiviral vector encoding Wiskott-Aldrich syndrome (WAS) protein
Period: Overall Study
Arm/Group | OTL-103 Gene Therapy
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: paediatric population
Arm/Group | OTL-103 Gene Therapy
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety of Reduced Conditioning Regimen
Description: The absence of prolonged aplasia (defined as ANC <0.5×10^9/L [<500/μL] at Day +60, with no evidence of BM recovery and requiring backup administration) was assumed as demonstrating the safety of the RIC regimen.
Time Frame: Follow up phase - Median duration: 11.1 years (range: 8.01 -13.3 years)
Population: Mobilization Set (MS) for Safety analysis. Intent-to-treat (ITT) population for Efficacy analysis. All eight enrolled participants were included in the ITT and MS populations
Measure: Count of Participants; unit: Participants
Arm/Group | TLT003 Gene Therapy
Number analyzed (Participants) | 8
Participants | 8

2. Primary Outcome: Safety of Lentivirus Gene Transfer Into HSC
Description: Safety and tolerability of lentiviral-transduced cell infusion. This will be evaluated on the basis of adverse events reporting and monitoring of the systemic reactions to cell infusion.
Time Frame: after 48 hours after Telethon003 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | TLT003 Gene Therapy
Number analyzed (Participants) | 8
Participants | 8

3. Primary Outcome: Sustained Engraftment of Genetically Corrected Haematopoietic Stem Cells in Peripheral Blood and/or in Bone Marrow
Description: Engraftment is characterized by the presence of gene modified cells in the BM or PB compartments. The main indicator of gene correction is detection of the WAS LVV sequences in the HSPCs and their progeny.
  The VCN, which is the mean number of integrated copies of the vector sequences per cell genome, was measured using PCR-based methods in DNA samples extracted from BM and PB cell populations at various timepoints post-treatment.
  Adequate engraftment was defined as either ≥0.04 VCN/cell in BM CD34+ cells or ≥0.01 VCN/cell in PB CD3+ cells.
Time Frame: at 1 year after Telethon003 infusion
Population: count of participants with sustained engraftment of genetically corrected HSPCs
Measure: Count of Participants; unit: Participants
Arm/Group | TLT003 Gene Therapy
Number analyzed (Participants) | 8
Participants | 8

4. Primary Outcome: Presence of Detectable Vector-derived WASP
Description: The percentage of subjects who present the proportion of PB cells expressing WASP was assessed by flow cytometry analysis.
Time Frame: Median duration: 11.1 years (range: 8.01 -13.3 years)
Measure: Count of Participants; unit: Participants
Arm/Group | TLT003 Gene Therapy
Number analyzed (Participants) | 8
Participants | 8

5. Primary Outcome: Improved T-cell Functions
Description: Improvement in in vitro T-cell proliferation was assessed upon stimulation with 3 doses of anti-immobilized CD3 (CD3i) monoclonal antibodies ≥1 year after Telethon003 infusion (as compared with pre-GT values) in PBMC and/or T-cell lines. The degree of correction was evaluated with respect to healthy controls.
Time Frame: Follow up phase - Median duration: 11.1 years (range: 8.01 -13.3 years)
Measure: Count of Participants; unit: Participants
Arm/Group | TLT003 Gene Therapy
Number analyzed (Participants) | 8
Participants | 8

6. Primary Outcome: Antigen-specific Responses to Vaccination
Description: The ability to mount a protective humoral response to at least 4 out of 5 nominal antigens including antibodies to T-cell dependent antigens and conjugated or unconjugated polysaccharide antigens was measured after vaccination (planned >1 year after Telethon003 infusion). If results were available on n <5 antigens, the rule of at least n-1 applied to define success.
Time Frame: Follow up phase - Median duration: 11.1 years (range: 8.01 -13.3 years)
Measure: Number; unit: participants
Arm/Group | TLT003 Gene Therapy
Number analyzed (Participants) | 8
participants | 7

7. Primary Outcome: Improved Platelet Count and MPV Normalization
Description: Sustained increase in platelet count compared to baseline, analyzing the individual longitudinal profile
Time Frame: up to 3 years after Telethon003 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | TLT003 Gene Therapy
Number analyzed (Participants) | 8
Participants | 8

8. Primary Outcome: Overall Survival
Description: Participant survival was monitored throughout the study.
Time Frame: Follow up phase - Median duration: 11.1 years (range: 8.01 -13.3 years)
Measure: Count of Participants; unit: Participants
Arm/Group | TLT003 Gene Therapy
Number analyzed (Participants) | 8
Participants | 8

9. Secondary Outcome: Lack of Immune Response to Transgene
Description: Anti-WASP and anti-HIV-1 antibodies (anti-p24) were monitored to evaluate response to transgene and to vector, respectively.
Time Frame: up to 3 years after Telethon003 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | TLT003 Gene Therapy
Number analyzed (Participants) | 8
Participants | 8

10. Secondary Outcome: Reduced Frequency of Severe Infections
Description: Decrease in number of severe infections as evaluated in the second and third year after the treatment by clinical history, complete physical examinations, hematological and microbiological tests.
Time Frame: up to 3 years after Telethon003 infusion
Reporting Status: Not Posted

11. Secondary Outcome: Reduced Bruising and Bleeding Episodes
Description: Reduction in bruising and/or bleeding manifestations when present, as assessed by clinical monitoring, compared to clinical history
Time Frame: 3 years
Reporting Status: Not Posted

12. Secondary Outcome: Reduced Autoimmunity Phenomena and Eczema
Description: Reduction in laboratory markers (number and titer of antibody when available) and/or clinical manifestations of autoimmunity, as evaluated by organ-specific and systemic autoantibodies, imaging and clinical follow-up, compared to clinical history. Reduction in eczema as evaluated by clinical score
Time Frame: 3 years
Reporting Status: Not Posted

13. Secondary Outcome: Improved Quality of Life
Description: Improved quality of life, measured after the first year of treatment by reduced hospitalization, reduced requirement of drugs, school attendance, social activities.
Time Frame: 3 year
Reporting Status: Not Posted

14. Secondary Outcome: Multilineage Engraftment of Genetically Corrected Cells
Description: ≥0.04 VCN/cell on all the available peripheral blood and/or bone marrow cell subpopulations (BM subpopulations: GlyA+, CD15+, CD61+, CD3+, CD19+, CD56+; PB subpopulations: CD15+, CD19+, CD56+)
Time Frame: 3 years
Reporting Status: Not Posted

15. Secondary Outcome: Overall Safety of the Treatment
Description: Recording of AE, AR, SAE/SAR, UAR, SUSAR
Time Frame: 8 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were reported in the statistical outputs from Screening onward. Post-treatment AEs were recorded during follow up - Median duration of follow-up was 11.1 (range: 8.0-13.3) years.
Description: For each AE, the Investigator specified the date of onset, intensity, action taken, corrective therapy given, outcome, assessment regarding the causal relationship with the IMP. Adverse events were graded according to the CTCAE scale. Events meeting the Hy's law criteria ( [ALT] ≥3×upper limit of normal [ULN] and bilirubin ≥2×ULN [>35% direct bilirubin] or ALT ≥3×ULN and international normalized ratio >1.5, if international normalized ratio measured) were to be reported as SAEs.
Arm/Group | OTL-103 Gene Therapy
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 8/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTL-103 Gene Therapy (N=8)
Mesenteric lymphadenitis (Blood and lymphatic system disorders) | 1 — Post-Treatment
Neutropenia (Blood and lymphatic system disorders) | 1 — Post-Treatment
Vomiting (Gastrointestinal disorders) | 1 — Post-Treatment
Pyrexia (General disorders) | 3 — Post-Treatment
Food Allergy (Immune system disorders) | 1 — Post-Treatment
Device related infection (Infections and infestations) | 2 — Post-Treatment
Gastroenteritis (Infections and infestations) | 1 — Post-Treatment
Pneumonia aspiration (Infections and infestations) | 1 — Post-Treatment
Appendicitis (Infections and infestations) | 1 — Post-Treatment
Aspergillus infection (Infections and infestations) | 1 — Post-Treatment
Bacterial sepsis (Infections and infestations) | 1 — Post-Treatment
Cellulitis (Infections and infestations) | 1 — Post-Treatment
Device related sepsis (Infections and infestations) | 1 — Post-Treatment
Gastroenteritis rotavirus (Infections and infestations) | 1 — Post-Treatment
Influenza (Infections and infestations) | 1 — Post-Treatment
Otitis media (Infections and infestations) | 1 — Post-Treatment
Pneumonia bacterial (Infections and infestations) | 1 — Post-Treatment
Tooth Abscess (Infections and infestations) | 1 — Post-Treatment
Tracheitis (Infections and infestations) | 1 — Post-Treatment
Viral infection (Infections and infestations) | 1 — Post-Treatment
Head injury (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 — Post-Treatment
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Post-Treatment
Irritability (Psychiatric disorders) | 1 — Post-Treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTL-103 Gene Therapy (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 — Post-Treatment
Eosinophilia (Blood and lymphatic system disorders) | 2 — Post-Treatment
Neutropenia (Blood and lymphatic system disorders) | 2 — Post-Treatment
Anaemia (Blood and lymphatic system disorders) | 2 — Post-Treatment
Febrile neutropenia (Blood and lymphatic system disorders) | 2 — Post-Treatment
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 — Post-Treatment
Polycythaemia (Blood and lymphatic system disorders) | 2 — Post-Treatment
Coagulopathy (Blood and lymphatic system disorders) | 1 — Post-Treatment
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 — Post-Treatment
Neutrophilia (Blood and lymphatic system disorders) | 1 — Post-Treatment
Splenomegaly (Blood and lymphatic system disorders) | 1 — Post-Treatment
Sinus tachycardia (Cardiac disorders) | 1 — Post-Treatment
Supraventricular extrasystoles (Cardiac disorders) | 1 — Post-Treatment
Phimosis (Congenital, familial and genetic disorders) | 3 — Post-Treatment
Familial mediterranean fever (Congenital, familial and genetic disorders) | 1 — Post-Treatment
Lymphatic malformation (Congenital, familial and genetic disorders) | 1 — Post-Treatment
Retinal anomaly congenital (Congenital, familial and genetic disorders) | 1 — Post-Treatment
Ear pain (Ear and labyrinth disorders) | 1 — Post-Treatment
Deafness neurosensory (Ear and labyrinth disorders) | 1 — Post-Treatment
Middle ear inflammation (Ear and labyrinth disorders) | 1 — Post-Treatment
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 — Post-Treatment
Adrenal insufficiency (Endocrine disorders) | 1 — Post-Treatment
Graves' disease (Endocrine disorders) | 1 — Post-Treatment
Hypoaldosteronism (Endocrine disorders) | 1 — Post-Treatment
Hypothyroidism (Endocrine disorders) | 1 — Post-Treatment
Precocious puberty (Endocrine disorders) | 1 — Post-Treatment
Eye inflammation (Eye disorders) | 3 — Post-Treatment
Conjunctivitis allergic (Eye disorders) | 2 — Post-Treatment
Blepharitis (Eye disorders) | 1 — Post-Treatment
Dyschromatopsia (Eye disorders) | 1 — Post-Treatment
Eczema eyelids (Eye disorders) | 1 — Post-Treatment
Astigmatism (Eye disorders) | 1 — Post-Treatment
Conjunctival haemorrhage (Eye disorders) | 1 — Post-Treatment
Conjunctival hyperaemia (Eye disorders) | 1 — Post-Treatment
Eyelid ptosis (Eye disorders) | 1 — Post-Treatment
Keratitis (Eye disorders) | 1 — Post-Treatment
Myopia (Eye disorders) | 1 — Post-Treatment
Periorbital oedema (Eye disorders) | 1 — Post-Treatment
Retinopathy (Eye disorders) | 1 — Post-Treatment
Visual acuity reduced (Eye disorders) | 1 — Post-Treatment
Diarrhoea (Gastrointestinal disorders) | 7 — Post-Treatment
Gingival bleeding (Gastrointestinal disorders) | 1 — Post-Treatment
Haematochezia (Gastrointestinal disorders) | 4 — Post-Treatment
Vomiting (Gastrointestinal disorders) | 3 — Post-Treatment
Dental caries (Gastrointestinal disorders) | 4 — Post-Treatment
Mouth haemorrhage (Gastrointestinal disorders) | 3 — Post-Treatment
Anal fissure (Gastrointestinal disorders) | 4 — Post-Treatment
Abdominal pain (Gastrointestinal disorders) | 2 — Post-Treatment
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 3 — Post-Treatment
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 — Post-Treatment
Malocclusion (Gastrointestinal disorders) | 4 — Post-Treatment
Aphthous ulcer (Gastrointestinal disorders) | 1 — Post-Treatment
Constipation (Gastrointestinal disorders) | 3 — Post-Treatment
Oral pain (Gastrointestinal disorders) | 2 — Post-Treatment
Stomatitis (Gastrointestinal disorders) | 2 — Post-Treatment
Tooth discolouration (Gastrointestinal disorders) | 2 — Post-Treatment
Anal haemorrhage (Gastrointestinal disorders) | 1 — Post-Treatment
Crohn's disease (Gastrointestinal disorders) | 1 — Post-Treatment
Dysphagia (Gastrointestinal disorders) | 1 — Post-Treatment
Enterocutaneous fistula (Gastrointestinal disorders) | 1 — Post-Treatment
Gastric disorder (Gastrointestinal disorders) | 1 — Post-Treatment
Gastric haemorrhage (Gastrointestinal disorders) | 1 — Post-Treatment
Gingival disorder (Gastrointestinal disorders) | 1 — Post-Treatment
Ileal ulcer (Gastrointestinal disorders) | 1 — Post-Treatment
Inguinal hernia (Gastrointestinal disorders) | 1 — Post-Treatment
Large intestinal ulcer (Gastrointestinal disorders) | 1 — Post-Treatment
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 — Post-Treatment
Oral disorder (Gastrointestinal disorders) | 1 — Post-Treatment
Pyrexia (General disorders) | 8 — Post-Treatment
Inflammation (General disorders) | 1 — Post-Treatment
Catheter site haemorrhage (General disorders) | 2 — Post-Treatment
Swelling face (General disorders) | 1 — Post-Treatment
Vaccination site inflammation (General disorders) | 2 — Post-Treatment
Catheter site erythema (General disorders) | 1 — Post-Treatment
Catheter site inflammation (General disorders) | 2 — Post-Treatment
Catheter site rash (General disorders) | 1 — Post-Treatment
Adverse drug reaction (General disorders) | 1 — Post-Treatment
Asthenia (General disorders) | 1 — Post-Treatment
Catheter site mass (General disorders) | 1 — Post-Treatment
Drug withdrawal syndrome (General disorders) | 1 — Post-Treatment
Feeling abnormal (General disorders) | 1 — Post-Treatment
Influenza like illness (General disorders) | 1 — Post-Treatment
Non-cardiac chest pain (General disorders) | 1 — Post-Treatment
Hepatomegaly (Hepatobiliary disorders) | 1 — Post-Treatment
Gallbladder disorder (Hepatobiliary disorders) | 1 — Post-Treatment
Hypertransaminasaemia (Hepatobiliary disorders) | 1 — Post-Treatment
Allergy to immunoglobulin therapy (Immune system disorders) | 3 — Post-Treatment
Food allergy (Immune system disorders) | 2 — Post-Treatment
Hypersensitivity (Immune system disorders) | 1 — Post-Treatment
Drug hypersensitivity (Immune system disorders) | 1 — Post-Treatment
Hypogammaglobulinaemia (Immune system disorders) | 1 — Post-Treatment
Upper respiratory tract infection (Infections and infestations) | 8 — Post-Treatment
Rhinitis (Infections and infestations) | 6 — Post-Treatment
Otitis media (Infections and infestations) | 3 — Post-Treatment
Otitis media acute (Infections and infestations) | 4 — Post-Treatment
Pharyngitis (Infections and infestations) | 4 — Post-Treatment
Conjunctivitis (Infections and infestations) | 4 — Post-Treatment
Gastroenteritis (Infections and infestations) | 3 — Post-Treatment
Ear infection (Infections and infestations) | 5 — Post-Treatment
Influenza (Infections and infestations) | 5 — Post-Treatment
Respiratory tract infection (Infections and infestations) | 4 — Post-Treatment
Sinusitis (Infections and infestations) | 4 — Post-Treatment
Cytomegalovirus infection reactivation (Infections and infestations) | 3 — Post-Treatment
Pneumonia (Infections and infestations) | 4 — Post-Treatment
Coronavirus infection (Infections and infestations) | 4 — Post-Treatment
Pharyngitis streptococcal (Infections and infestations) | 1 — Post-Treatment
Skin infection (Infections and infestations) | 2 — Post-Treatment
Tooth abscess (Infections and infestations) | 2 — Post-Treatment
Eye infection (Infections and infestations) | 3 — Post-Treatment
Amoebic dysentery (Infections and infestations) | 1 — Post-Treatment
Bacterial disease carrier (Infections and infestations) | 1 — Post-Treatment
Catheter site infection (Infections and infestations) | 2 — Post-Treatment
Diarrhoea infectious (Infections and infestations) | 2 — Post-Treatment
Folliculitis (Infections and infestations) | 1 — Post-Treatment
Nasopharyngitis (Infections and infestations) | 3 — Post-Treatment
Oral candidiasis (Infections and infestations) | 3 — Post-Treatment
Oral herpes (Infections and infestations) | 1 — Post-Treatment
Tracheitis (Infections and infestations) | 1 — Post-Treatment
Urinary tract infection (Infections and infestations) | 1 — Post-Treatment
Viral infection (Infections and infestations) | 2 — Post-Treatment
Abscess limb (Infections and infestations) | 1 — Post-Treatment
Bronchitis (Infections and infestations) | 2 — Post-Treatment
COVID-19 (Infections and infestations) | 2 — Post-Treatment
Cytomegalovirus infection (Infections and infestations) | 1 — Post-Treatment
Cytomegalovirus viraemia (Infections and infestations) | 1 — Post-Treatment
Epstein-Barr virus infection (Infections and infestations) | 2 — Post-Treatment
Escherichia urinary tract infection (Infections and infestations) | 2 — Post-Treatment
Gastroenteritis viral (Infections and infestations) | 2 — Post-Treatment
Paronychia (Infections and infestations) | 1 — Post-Treatment
Pharyngotonsillitis (Infections and infestations) | 1 — Post-Treatment
Urethritis (Infections and infestations) | 1 — Post-Treatment
Urinary tract infection bacterial (Infections and infestations) | 1 — Post-Treatment
Viral rhinits (Infections and infestations) | 1 — Post-Treatment
Amoebiasis (Infections and infestations) | 1 — Post-Treatment
Bordetella infection (Infections and infestations) | 1 — Post-Treatment
Chronic tonisllitis (Infections and infestations) | 1 — Post-Treatment
Conjunctivitis bacterial (Infections and infestations) | 1 — Post-Treatment
Coxsackie vital infection (Infections and infestations) | 1 — Post-Treatment
Ear infection fungal (Infections and infestations) | 1 — Post-Treatment
Enterobiasis (Infections and infestations) | 1 — Post-Treatment
Enterococcal sepsis (Infections and infestations) | 1 — Post-Treatment
Enterocolitis viral (Infections and infestations) | 1 — Post-Treatment
Fungal skin infection (Infections and infestations) | 1 — Post-Treatment
Genital infection fungal (Infections and infestations) | 1 — Post-Treatment
Gingivitis (Infections and infestations) | 1 — Post-Treatment
Herpes virus infection (Infections and infestations) | 1 — Post-Treatment
Infection parasitic (Infections and infestations) | 1 — Post-Treatment
Laryngitis (Infections and infestations) | 1 — Post-Treatment
Laryngopharyngitis (Infections and infestations) | 1 — Post-Treatment
Lice infestation (Infections and infestations) | 1 — Post-Treatment
Measles (Infections and infestations) | 1 — Post-Treatment
Molluscum contagiosum (Infections and infestations) | 1 — Post-Treatment
Omphalitis (Infections and infestations) | 1 — Post-Treatment
Otitis externa (Infections and infestations) | 1 — Post-Treatment
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 — Post-Treatment
Pneumonia cytomegaloviral (Infections and infestations) | 1 — Post-Treatment
Pulpitis dental (Infections and infestations) | 1 — Post-Treatment
Respiratory tract infection viral (Infections and infestations) | 1 — Post-Treatment
Varicella (Infections and infestations) | 1 — Post-Treatment
Viral upper respiratory tract infection (Infections and infestations) | 1 — Post-Treatment
Head injury (Injury, poisoning and procedural complications) | 3 — Post-Treatment
Limb injury (Injury, poisoning and procedural complications) | 4 — Post-Treatment
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 — Post-Treatment
Face injury (Injury, poisoning and procedural complications) | 2 — Post-Treatment
Hand fracture (Injury, poisoning and procedural complications) | 2 — Post-Treatment
Torus fracture (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Ankle fracture (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Arthropod bite (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Eyelid injury (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Fall (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Infusion related reaction (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Joint injury (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Lip injury (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Tibia fracture (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Vaccination complication (Injury, poisoning and procedural complications) | 1 — Post-Treatment
Anti-platelet antibody positive (Investigations) | 8 — Post-Treatment
Staphylococcus test positive (Investigations) | 5 — Post-Treatment
Hepatic enzyme increased (Investigations) | 3 — Post-Treatment
Antineutrophil cytoplasmic antibody positive (Investigations) | 5 — Post-Treatment
Streptococcus test positive (Investigations) | 4 — Post-Treatment
Antinuclear antibody positive (Investigations) | 3 — Post-Treatment
Blood immunoglonulin E increased (Investigations) | 4 — Post-Treatment
Blood alkaline phosphatase increased (Investigations) | 3 — Post-Treatment
Cytomegalovirus test positive (Investigations) | 2 — Post-Treatment
Haemophilus test positive (Investigations) | 3 — Post-Treatment
Pseudomonas test positive (Investigations) | 1 — Post-Treatment
Smooth muscle antibody positive (Investigations) | 3 — Post-Treatment
Vitamin D decreased (Investigations) | 3 — Post-Treatment
Blood calcium decreased (Investigations) | 2 — Post-Treatment
Clostridium test positive (Investigations) | 2 — Post-Treatment
Electrophoresis protein abnormal (Investigations) | 2 — Post-Treatment
Intraocular pressure increased (Investigations) | 1 — Post-Treatment
Adenovirus test positive (Investigations) | 2 — Post-Treatment
Anti-saccharomyces cerevisiae antibody test positive (Investigations) | 2 — Post-Treatment
C-reactive protein increased (Investigations) | 1 — Post-Treatment
Coombs direct test positive (Investigations) | 1 — Post-Treatment
Epstein-Barr virus test positive (Investigations) | 1 — Post-Treatment
Inflammatory marker increased (Investigations) | 1 — Post-Treatment
Serum ferritin decreased (Investigations) | 2 — Post-Treatment
Serum ferritin increased (Investigations) | 1 — Post-Treatment
Acinetobacter test positive (Investigations) | 1 — Post-Treatment
Anti-thyroid antibody positive (Investigations) | 1 — Post-Treatment
Anti-transglutaminase antibody increased (Investigations) | 1 — Post-Treatment
Antimitochondrial antibody positive (Investigations) | 1 — Post-Treatment
Antiribosomal P antibody positive (Investigations) | 1 — Post-Treatment
Aspartate aminotransferase increased (Investigations) | 1 — Post-Treatment
Blood beta-D-glucan abnormal (Investigations) | 1 — Post-Treatment
Blood bicarbonate decreased (Investigations) | 1 — Post-Treatment
Blood bilirubin increased (Investigations) | 1 — Post-Treatment
Blood cholesterol increased (Investigations) | 1 — Post-Treatment
Blood creatinine increased (Investigations) | 1 — Post-Treatment
Blood culture positive (Investigations) | 1 — Post-Treatment
Blood folate decreased (Investigations) | 1 — Post-Treatment
Blood glucose increased (Investigations) | 1 — Post-Treatment
Blood iron decreased (Investigations) | 1 — Post-Treatment
Blood thyroid stimulating hormone increased (Investigations) | 1 — Post-Treatment
Candida test positive (Investigations) | 1 — Post-Treatment
Chest X-ray abnormal (Investigations) | 1 — Post-Treatment
Dehydroepiandrosterone decreased (Investigations) | 1 — Post-Treatment
Double stranded DNA antibody positive (Investigations) | 1 — Post-Treatment
Enterobacter test positive (Investigations) | 1 — Post-Treatment
Faecal calprotectin increased (Investigations) | 1 — Post-Treatment
Lymph nodes scan abnormal (Investigations) | 1 — Post-Treatment
Moraxella test positive (Investigations) | 1 — Post-Treatment
Occult blood (Investigations) | 1 — Post-Treatment
Spirometry abnormal (Investigations) | 1 — Post-Treatment
Transaminases increased (Investigations) | 1 — Post-Treatment
Tri-iodothyronine increased (Investigations) | 1 — Post-Treatment
Vitamin B12 increased (Investigations) | 1 — Post-Treatment
Hypokalaemia (Metabolism and nutrition disorders) | 6 — Post-Treatment
Iron deficiency (Metabolism and nutrition disorders) | 5 — Post-Treatment
Obesity (Metabolism and nutrition disorders) | 1 — Post-Treatment
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 — Post-Treatment
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 — Post-Treatment
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 — Post-Treatment
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 — Post-Treatment
Hyponatraemia (Metabolism and nutrition disorders) | 1 — Post-Treatment
Insulin resistance (Metabolism and nutrition disorders) | 2 — Post-Treatment
Feeding intolerance (Metabolism and nutrition disorders) | 1 — Post-Treatment
Hyperglycaemia (Metabolism and nutrition disorders) | 1 — Post-Treatment
Hyperkalaemia (Metabolism and nutrition disorders) | 1 — Post-Treatment
Weight gain poor (Metabolism and nutrition disorders) | 1 — Post-Treatment
Arthritis (Musculoskeletal and connective tissue disorders) | 1 — Post-Treatment
Osteitis (Musculoskeletal and connective tissue disorders) | 1 — Post-Treatment
Back pain (Musculoskeletal and connective tissue disorders) | 3 — Post-Treatment
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 — Post-Treatment
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 — Post-Treatment
Short stature (Musculoskeletal and connective tissue disorders) | 1 — Post-Treatment
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 — Post-Treatment
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Post-Treatment
Headache (Nervous system disorders) | 3 — Post-Treatment
Cerebral cyst (Nervous system disorders) | 1 — Post-Treatment
Dyskinesia (Nervous system disorders) | 1 — Post-Treatment
Speech disorder (Nervous system disorders) | 1 — Post-Treatment
Aggression (Psychiatric disorders) | 1 — Post-Treatment
Anxiety (Psychiatric disorders) | 1 — Post-Treatment
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 — Post-Treatment
Autism spectrum disorder (Psychiatric disorders) | 1 — Post-Treatment
Behaviour disorder (Psychiatric disorders) | 1 — Post-Treatment
Depression (Psychiatric disorders) | 1 — Post-Treatment
Drug dependece (Psychiatric disorders) | 1 — Post-Treatment
Enuresis (Psychiatric disorders) | 1 — Post-Treatment
Sleep disorder (Psychiatric disorders) | 1 — Post-Treatment
Haematuria (Renal and urinary disorders) | 1 — Post-Treatment
Proteinuria (Renal and urinary disorders) | 1 — Post-Treatment
Pyelocaliectasis (Renal and urinary disorders) | 2 — Post-Treatment
Acute kidney injury (Renal and urinary disorders) | 1 — Post-Treatment
Nephrolothiasis (Renal and urinary disorders) | 1 — Post-Treatment
Pollakiuria (Renal and urinary disorders) | 1 — Post-Treatment
Polyuria (Renal and urinary disorders) | 1 — Post-Treatment
Renal impairment (Renal and urinary disorders) | 1 — Post-Treatment
Balanoposthitis (Reproductive system and breast disorders) | 3 — Post-Treatment
Acquired phimosis (Reproductive system and breast disorders) | 2 — Post-Treatment
Penile erythema (Reproductive system and breast disorders) | 1 — Post-Treatment
Perineal erythema (Reproductive system and breast disorders) | 1 — Post-Treatment
Varicocele (Reproductive system and breast disorders) | 1 — Post-Treatment
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 — Post-Treatment
Cough (Respiratory, thoracic and mediastinal disorders) | 5 — Post-Treatment
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 — Post-Treatment
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 — Post-Treatment
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 — Post-Treatment
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 — Post-Treatment
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 — Post-Treatment
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 — Post-Treatment
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 — Post-Treatment
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 — Post-Treatment
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Nasal varices (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 — Post-Treatment
Petechiae (Skin and subcutaneous tissue disorders) | 7 — Post-Treatment
Eczema (Skin and subcutaneous tissue disorders) | 6 — Post-Treatment
Rash (Skin and subcutaneous tissue disorders) | 4 — Post-Treatment
Drug eruption (Skin and subcutaneous tissue disorders) | 3 — Post-Treatment
Dermatitis (Skin and subcutaneous tissue disorders) | 4 — Post-Treatment
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 — Post-Treatment
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 — Post-Treatment
Urticaria (Skin and subcutaneous tissue disorders) | 2 — Post-Treatment
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 — Post-Treatment
Pruritus (Skin and subcutaneous tissue disorders) | 2 — Post-Treatment
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 — Post-Treatment
Erythema (Skin and subcutaneous tissue disorders) | 2 — Post-Treatment
Pityriasis alba (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Dry skin (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Purpura (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Skin fissures (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Skin lesion (Skin and subcutaneous tissue disorders) | 1 — Post-Treatment
Vasculitis (Vascular disorders) | 1 — Post-Treatment
Hypertension (Vascular disorders) | 1 — Post-Treatment
Phlebitis (Vascular disorders) | 2 — Post-Treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall send any manuscript to the Sponsor/FT prior to its submission for publication. The Sponsor/FT shall have 45 days (silence=consent), from receipt of the manuscript, during which time any manuscript amendments may be suggested. The Principal Investigator shall accept the incorporation into the publication of any comments that do not affect the reliability of data, as well as the rights, safety and well-being of the patients.

DOCUMENTS (2):
  • Study Protocol (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT01515462/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT01515462/SAP_001.pdf